CLINICAL TRIAL: NCT01205243
Title: An Open Label, Multi-centre, Non-interventional Post-marketing Surveillance (PMS) to Monitor the Safety and Efficacy of ZIAGEN® Administered in Korean Patients According to the Prescribing Information
Brief Title: ZIAGEN® Post-marketing Surveillance
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114382
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Infection, Human Immunodeficiency Virus I
Keywords: Abacavir; post-marketing surveillance
MeSH Terms: conditions — Infections | interventions — abacavir

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ZIAGEN®: Patients administrated ZIAGEN® at the site
  Interventions: Drug: ZIAGEN®

INTERVENTIONS:
Drug: ZIAGEN® — Basically there is no treatment allocation. Subjects who would be administrated ZIAGEN® at their physician's discretion will be enrolled. Dosage regimen will be recommended according to the prescribing information. Subjects will be enrolled consecutively.

SUMMARY:
An open label, multi-centre, non-interventional post-marketing surveillance (PMS) to monitor the safety and efficacy of ZIAGEN® administered in Korean patients according to the prescribing information.

DETAILED DESCRIPTION:
This study will collect clinical data, mainly focused on safety, in Korean population as per the requirement of KFDA for market authorization.

ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship.

ELIGIBILITY:
All subjects must satisfy the following criteria.

* Subject who is treated in combination with other antiretroviral agents for the treatment of HIV infection.
* Subject who is considered to follow this post marketing surveillance protocol by the investigator.
* Subject who is treated with ZIAGEN® according to the prescribing information. As considering the characteristic of observational post marketing surveillance, the exclusion criteria is not strict. All investigators should prescribe ZIAGEN® according to the prescribing information which approved in Korea.
* Subjects with hypersensitivity to ZIAGEN® or ingredients
* Subjects with moderate or severe hepatic impairment
* Subject with end-stage renal disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients administrated ZIAGEN® at the site
Sampling Method: Probability Sample
Enrollment: 671 (Actual)
Dates: Start 2010-11-01; Primary Completion 2015-02-01 (Actual); Study Completion 2015-02-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse event after ZIAGEN® administration | 12month

SECONDARY OUTCOMES:
Occurrence of serious adverse event after ZIAGEN® administration | 12month
efficacy after ZIAGEN® administration | 12month
Occurrence of unexpected adverse drug reaction after ZIAGEN® administration | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Incheon, South Korea